CLINICAL TRIAL: NCT06675097
Title: Assessment of the Impact of Intestinal Gas Emission Quality on the Postoperative Course After Abdominal Surgery: Single-center Prospective Study - FLATQUAL- Abdominal Surgery and Gas Transit
Brief Title: Assessment of the Impact of Intestinal Gas Emission Quality on the Postoperative Course After Abdominal Surgery
Acronym: FLATQUAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0335
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Complication; Recovery, Physiological
Keywords: transit; surgery; abdomen; stool; gas
MeSH Terms: conditions — Postoperative Complications; Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recovery of transit after surgery is an important parameter in postoperative evaluation. It generally reflects simple postoperative outcomes and allows the patient to return home.

The quality of gas recovery after surgery has not been studied to our knowledge, but it is not uncommon for an operated patient to emit some gas considered as a recovery of transit when it is ultimately a false transit preceding a postoperative ileus. Furthermore, intestinal gases and their composition reflect the intestinal microbiota. This microbiota has been shown to be predictive of the appearance of an operative complication. As the analysis of this microbiota cannot be carried out routinely, it is important to be able to use a reflection of this microbiota in routine practice and to correlate it with the surgical outcomes. Intestinal gas therefore seems to be the tool of choice.

The main objective is to evaluate the association between the appearance of an operative complication and the resumption of gas transit qualified according to its quantity and quality.

The secondary objectives are to compare the quantity and quality of gases pre- and post-operatively and to define a predictive score for surgical complications, based on the number and quality of post-surgical gases.

Data regarding gas transit are collected by the patient in a questionnaire the two days before the surgery and until the patient leaves hospital (or until day 15 post-operative if the patient is still hospitalized).

Data regarding possible complications ((defined according to Dindo-Clavien as any deviation from the expected postoperative outcomes within 90 days following surgery) are collected throughout the hospital stay (day 0 : surgery to day 15 post-operatively), during the post-operative consultation (day 30) and during a telephone call to the patient (day 90).

The expected results are to highlight a correlation between the quality/quantity of gases and post-operative outcomes. A predictive score for complications could then be proposed and validated during this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Indication for open or laparoscopic abdominal surgery
* Whose expected length of stay is ≥ 2 days

Non Inclusion Criteria:

* Patients requiring a stomy on the initial surgery
* Need for immediate postoperative intensive care
* Emergency surgery
* Patient not knowing how to read or write
* Poor understanding of the French language
* Person deprived of liberty by judicial or administrative decision
* Person subject to psychiatric care under duress
* Person subject to a legal protection measure
* Person unable to express consent
* Person objecting to participating in research

Exclusion Criteria:

-Immediate post-operative intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be included in the hospital they will be operated on
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association between the appearance of an operative complication and the resumption of gas transit qualified according to its quantity and quality. | From Day 0 (surgery) to the 90 post-operative days +/- 15 days.
  Operative complication is defined according to Dindo-Clavien as any deviation from the expected postoperative outcomes within 90 days following surgery. Complications are then classified according to the Dindo-Clavien classification from 1 (simplest) to 5 (death).
To evaluate the association between the appearance of an operative complication and the resumption of gas transit qualified according to its quantity and quality. | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized.From Day 0 (surgery) to the 90 post-operative days +/- 15 days.
  The resumption of gas transit will be defined as the emission of gas for at least 2 days in a row.
  • The quantity corresponds to the number / 24 hours of gas
To evaluate the association between the appearance of an operative complication and the resumption of gas transit qualified according to its quantity and quality. | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized.From Day 0 (surgery) to the 90 post-operative days +/- 15 days
  The resumption of gas transit will be defined as the emission of gas for at least 2 days in a row.
  • The quality is defined by:
  * Single or multiple over the same time
  * Noisy or soundless
  * Dry or wet (no stools but mucus or transparent liquids)
  * Accompanied by stools
  * Non-odorous, slightly odorous, very smelly
  * Painful before the show
  * Relief after emission

SECONDARY OUTCOMES:
to compare the quantity of gas pre- and post-operative | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized
  • gas quantity corresponds to number/24 H of gas (data are daily collected by the patient in a questionnaire)
to compare the quantity of stools pre- and post-operative | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized
  • Stoll quantity corresponds to number/24 H of stool (data are daily collected by the patient in a questionnaire)
to compare the quality of gases pre- and post-operative | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized
  • Gas quality is defined by :
  * Single or multiple over the same time
  * Noisy or soundless
  * Dry or wet (no stools but mucus or transparent liquids)
  * Accompanied by stools
  * Non-odorous, slightly odorous, very smelly
  * Painful before the show
  * Relief after emission
  .Data from gas are daily collected by the patient in a questionnaire.
to compare the quality of stool pre- and post-operative | The 2 days before surgery and up to 15 days post-operative if the patient is still hospitalized
  •stool quality is defined by the Bristol scale (type 1: separate hard lumps (severe constipation); type 2: lumpy and sausage-like (mild constipation); type 3: sausage shape with cracks (normal); type 5: soft blobs with clear-cut edges (lacking fiber); type 6: mushy consistency with ragged edges (mild diarrhea); type 7: liquid consistency with no solid pieces (severe diarrhea).
  .data are daily collected by the patient in a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Angers Hospital (visceral surgery department), Angers, France

IPD SHARING:
Plan to Share IPD: No